CLINICAL TRIAL: NCT06773988
Title: Follow-up of NIV At Home in Patients with Duchenne Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68844
Record Dates: First submitted 2024-12-04; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; Non-invasive ventilation; Feasibility; Home unattended full-video polysomnography; Transcutaneous capnography
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with Duchenne using NIV in follow-up at the Leuven University Center for Sleep/wake: Patients with Duchenne Muscular Dystrophy (DMD) on non-invasive ventilation (NIV) who need a yearly follow up by polysomnopgraphy
  Interventions: Diagnostic Test: Monitoring of NIV at home

INTERVENTIONS:
Diagnostic Test: Monitoring of NIV at home — Monitoring of NIV at home

SUMMARY:
The aim of this study is to verify whether full video home polysomnography (sleep study) with nocturnal transcutaneous CO2 monitoring is feasible in the follow-up of non-invasive ventilation (NIV) in patients with Duchenne muscular dystrophy. The researchers would like to investigate whether they could perform sufficient measurements in the home situation and see if correct decision for further treatment could be made. Furthermore, the researchers will make an analysis on the minimal requirements of measurements to make a correct decision for the treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DMD > 18 years using NIV
* Signing the written informed consent

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are in follow-up at the Leuven University City for Sleep/wake disorders
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility of full video home polysomnography (PSG) and follow-up at home in patients with DMD on NIV, identical to the sophisticated PSG in-hospital | Yearly home polysomnopraphy and Transcutaneous CO2 measurement, for a period of 3 years
  The primary endpoint is the feasibility of a home based full-video polysomnography for follow-up of DMD patients on NIV.

SECONDARY OUTCOMES:
Analysis of the minimal equipment to assure a correct follow-up of NIV at home (full video PSG vs PtcCO2) measurement combined with ventilator software data vs ventilator software data vs PtcCO2 measurement) | 3 years
Cost-benefit analysis of follow-up of NIV at home as a preparation to create a file for the Belgian health insurance (registration of time and material) | Cost-benifit analysis will be carried out at study completion, after 3 years.
  During 3 years, the costs for performing a home based full-video PSG (relocation costs, material, physiotherapist wage) will be weighed against the benifits (patient comfort, relieving hospital ward occupation)
Amount of technical failures, i.e. PSG signals, PtcCO2 measurement, O2 saturation measurement and video monitoring. | Performed immediately after each PSG or PtcCO2 measurement, during a period of 3 years.
  Checklist after each PSG
Patient Reported Outcomes: Experience between in-hospital PSG vs PSG at home | The PROM will be completed by the patient at each yearly PSG, during the 3 years of the ongoing study
  Both patient and caregiver report on a 10 point likert scale, ranging from totally not to very, how mor comfortable the PSG at home was compared to the hospital PSG.
Sleep quality questionnaire: The Pittsburgh Sleep Quality Index (PSQI) | The PSQI will be completed by the patient at each yearly PSG and at each yearly PtcCO2 measurment, during 3 years.
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Home-NIV PROM: S3-NIV | The S3-NIV questionnaire will be completed by the patient at each yearly PSG and at each yearly PTCO2 measurement, during 3 years.
  The S3-NIV questionnaire is a short, valid and repeatable self-completed tool for the routine clinical assessment of patients undergoing home NIV. The S3-NIV questionnaire provides clinicians and patients with a simple and reliable tool to assess important domains (symptoms, sleep quality and NIV-related side effects) as a complement to physiological monitoring. The S3-NIV questionnaire has 11 items. Each item is scored using a 5-point Likert scale from "always true" to "never true". The total score and the two sub scores range from 0 to 10 points. Lower scores represent a higher, negative impact of the disease and NIV on the individual.
Daytime sleepiness questionnaire: Epworth Sleepiness Scale (ESS) | The ESS questionnaire will be completed by the patient at each yearly PSG and each yearly PtcCO2 measurement, during 3 years.
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruyneel M, Ninane V. Unattended home-based polysomnography for sleep disordered breathing: current concepts and perspectives. Sleep Med Rev. 2014 Aug;18(4):341-7. doi: 10.1016/j.smrv.2013.12.002. Epub 2013 Dec 12. PMID 24388970
- [Background] Toussaint M, Chatwin M, Soudon P. Mechanical ventilation in Duchenne patients with chronic respiratory insufficiency: clinical implications of 20 years published experience. Chron Respir Dis. 2007;4(3):167-77. doi: 10.1177/1479972307080697. PMID 17711917
- [Background] Bourke SC. Respiratory involvement in neuromuscular disease. Clin Med (Lond). 2014 Feb;14(1):72-5. doi: 10.7861/clinmedicine.14-1-72. No abstract available. PMID 24532751